CLINICAL TRIAL: NCT04098900
Title: Clinical Evaluation of the Click Sexual Health Test for the Detection of Neisseria Gonorrhoeae (NG), Trichomonas Vaginalis (TV), and Chlamydia Trachomatis (CT) in Women
Status: Completed | Type: Observational
Sponsor: Visby Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-000279
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-09

CONDITIONS: Chlamydial Infection; Gonococcal Infection; Trichomoniasis
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Trichomonas Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Click Sexual Health Test — The Click Device is a single-use (disposable), fully integrated, rapid, compact, device containing a polymerase chain reaction (PCR)-based nucleic acid amplification test (NAAT) for accurate, qualitative detection and differentiation of deoxyribonucleic acid (DNA) for Neisseria gonorrhea (NG), Trichomonas vaginalis (TV), and Chlamydia trachomatis (CT) organisms.

SUMMARY:
This study is a multi-center study with a minimum of three CLIA-waived intended operator sites in the United States in which prospectively self-collected vaginal specimens obtained from subjects who are symptomatic or asymptomatic for CT, NG, or TV will be evaluated with the Click Sexual Health Test in a Clinical Laboratory Improvement Amendments (CLIA) waived setting. Subjects interested in participating in this study will be assessed for eligibility and asked to give informed consent and assent, if applicable, by the Investigational Review Board (IRB). Only those subjects who meet the inclusion and exclusion criteria may be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give voluntary written informed consent and assent form (or the parental/legal guardian will provide parental permission) before any study-related procedure is performed.
2. Female at birth. (Pregnant and breastfeeding women are eligible).
3. Age greater than or equal to 14 years at the time of enrollment
4. Able to read and understand the procedural information provided for the study.
5. Able and willing to follow all study procedures, including performing self-collection of one vaginal swab and permitting a HCP to collect three additional vaginal swabs.

Exclusion Criteria:

1. Have a medical condition, serious intercurrent illness, or other circumstance that, in the Investigator's judgement, could jeopardize the subjects's safety, or could interfere with study procedures.
2. Enrollment in the DMID 18-0024 and this study previously.
3. Use of antiperspirants and deodorants or the following vaginal products: douches, washes, lubricants, vaginal wipes, vaginal moisturizers, or feminine hygiene spray in the genital area, within 48 hours prior to enrollment.

Ages: 14 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises female subjects greater than or equal to 14 years of age visiting any of the participating clinics for any reason, who may be symptomatic or asymptomatic for STIs at locations including but not limited to: OB/GYN and primary care offices, as well as sexually transmitted disease, teen, public health, and family planning clinics. Any subject who meets the inclusion/exclusion criteria is eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
The percent sensitivity and specificity of the Click Device for detection of CT in self-collected vaginal specimens as compared to Patient Infected Status (PIS) using vaginal specimens collected by a qualified Health Care Provider (HCP) | up to 6 months
The percent sensitivity and specificity of the Click Device for detection of NG in self-collected vaginal specimens as compared to PIS using vaginal specimens collected by a qualified HCP | up to 6 months
The percent sensitivity and specificity of the Click Device for detection of TV in self-collected vaginal specimens as compared to PIS using vaginal specimens collected by a qualified HCP | up to 6 months

SECONDARY OUTCOMES:
Usability will be measured by 5-point Likert scale responses, yes/no questions, and open text questions from study operators. | up to 6 months
  Questions are around three domains of interest: i) instructions, ii) operations, and iii) visual interpretation for the Click device for detection of CT, NG, and TV with patient self-collected specimens.
  The 5-point Likert scale will measure responses to questions in the form of: (1) Strongly Disagree, (2) Disagree, (3) Neutral, (4) Agree, and (5) Strongly Agree

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Planned Parenthood North Central States, Saint Paul, Minnesota
  - Planned Parenthood of the St. Louis Region and Southwest Missouri, St Louis, Missouri
  - Lawrence OB/GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Planned Parenthood Gulf Coast, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided